CLINICAL TRIAL: NCT02008045
Title: Advanced MR Imaging of Perinatal Brain Injury: Correlation With Neurocognitive Outcome
Brief Title: MR Imaging of Perinatal Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rafael Ceschin, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY19100215
Record Dates: First submitted 2013-11-15; First posted 2013-12-11 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Perinatal White Matter Brain Injury
Keywords: MRI; Imaging; Neurocognitive; White matter injury
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neonates at Risk for Brian Injury: Magnetic Resonance Imaging Neurodevelopmental Testing - 18 Month
  Interventions: Device: Magnetic Resonance Imaging; Behavioral: Neurodevelopmental Testing
- Term Neonates: Magnetic Resonance Imaging Neurodevelopmental Testing - 18 Month
  Interventions: Device: Magnetic Resonance Imaging; Behavioral: Neurodevelopmental Testing

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Brain MRI without Contrast
Behavioral: Neurodevelopmental Testing — Validated battery of neurodevelopmental and psychological tests.

SUMMARY:
The purpose of this study is to collect and compare information from cranial ultrasounds, magnetic resonance imaging scans, neurological exam and neuropsychological assessments of children. The investigators hope that the information collected in this study will help with early screening, diagnosis and treatment of brain injury in newborns as well as identify a connection between MR imaging (MRI-magnetic resonance imaging, MRS-magnetic resonance spectroscopy) and neurodevelopmental outcome.

DETAILED DESCRIPTION:
In the last two decades, major advances have been made in the clinical care of premature and term infants, including in the management of sepsis and respiratory compromise that can contribute to neurological disabilities in survivors. The incidence of classic cystic periventricular leukomalacia (PVL) has declined and a more diffuse and non-cystic pattern of cerebral white matter injury is more predominant. Although multiple pathologies occur in premature infants, the principal variety accounting for the predominance of neurodevelopmental disability is PVL. This disability in very low birth weight infants (VLBW) (< 1500 grams) includes cognitive/behavioral deficits in 25-50% and cerebral palsy in 5-10%. Neuroimaging studies of VLBW survivors suggest that the cerebral palsy is related to the focal necrotic lesions of PVL, whereas the cognitive/behavioral deficits correlate with more diffuse cerebral white matter injury. PVL is defined as damaged immature cerebral white matter with periventricular focal necrosis ("focal" component) in association with diffuse reactive gliosis and microglial activation in the surrounding white matter ("diffuse" component). Of note, PVL occurs in the late preterm infant and the term infant, particularly in cases of congenital heart disease. The pathogenesis of perinatal white matter injury is currently thought to be related to a complex interaction between maternal/fetal infection, cytokines and hypoxia-ischemia which results in both the generation of reactive oxygen specific agents (oxidative stress), apoptotic oligodendrocyte cell death, and axonal injury. In long-term survivors with PVL, neuroimaging studies often demonstrate reduced cerebral white matter volume, impaired myelination, ventriculomegaly and reduced volume in the cerebral cortex, thalamus/basal ganglia and cerebellum. In many of these long-term studies, the preterm children studies had normal cranial ultrasound. Cranial ultrasound, however, is not adequate for assessing non-cystic focal or diffuse white matter injury. To date, there are no longitudinal MR studies of preterm or congenital heart disease infants which correlate advanced neonatal MR imaging techniques with long-term neurodevelopmental outcome or advanced MR techniques performed in the childhood period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies and neonates with congenital heart disease
* Term Neonates

Exclusion Criteria:

* Severe congenital brain malformation
* Significant chromosomal abnormality / syndrome which could confound the neurodevelopmental follow up data
* Preterm birth and congenital heart disease
* Focal neurological abnormality
* Chronic seizures
* Severe congenital brain malformation
* Significant chromosomal abnormality/ syndrome which could confound the neurodevelopmental follow up data
* Major pregnancy complication (diabetes, eclampsia)
* Sepsis
* ECMO
* Significant birth trauma and/or hypoxic ischemic injury

Ages: 1 Day to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be enrolled between birth and 7 years of age.
Sampling Method: Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Developmental Assessment | 18 Months
  Administration of neurodevelopmental testing and completion of parent questionnaires regarding the child's development.

SECONDARY OUTCOMES:
Assessment of White Matter Injury in Brain | Baseline
  MR Scan
Changes in White Matter Injury from Baseline | at 6 Years
  MR Scan

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Panigrahy, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Materials generated under the project will be disseminated in accordance with the University of Pittsburgh and NIH policies. Depending on such policies, materials may be transferred to others under the terms of a material transfer agreement.
  Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. Research data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.
Time Frame: De-identified data will be shared once all study subjects have completed participation and data analysis has been completed.
Access Criteria: De-identified data will be shared via secure website with access granted by PI research team.